CLINICAL TRIAL: NCT02330055
Title: Determination of the Predictors of Nocturnal Desaturation in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Eikermann, MD PhD, Director of Research, Critical Care Division, Associate Professor of Anesthesia, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011P001326B
Record Dates: First submitted 2014-12-23; First posted 2015-01-01 (Estimated); Results first posted 2018-04-09 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Sleep Disordered Breathing; Nocturnal Oxygen Desaturation; Upper Airway Edema
MeSH Terms: conditions — Sleep Apnea Syndromes

ARMS (2):
- Forty-five degrees elevated upper body position (Active Comparator): If the patient is randomized in this study arm after enrollment, the investigators will elevate the patients upper body to 45 degree prior to sleeping. The patient will wear a pulseoximeter (WristOx Model 3150) during the night. The investigators will collect the SpO2 and pulse rate with this device and then quantify desaturation events.
  The investigators will ask the patient to fill out a questionnaire, which includes the P-SAP score, the STOP-BANG score, the Epworth Sleepiness Scale and the self-reported pain.
  Interventions: Procedure: Forty-five degrees elevated upper body position; Device: Noninvasive wrist pulse oximeter (WristOx Model 3150); Other: Stop-Bang questionnaire; Other: Epworth Sleepiness Scale; Other: P-SAP Score; Other: self-reported pain
- Non-elevated upper body position (Placebo Comparator): If the patient is randomized in this study arm after enrollment, the investigators will flatten the patients upper body to a supine position prior to sleeping. The patient will wear a pulseoximeter (WristOx Model 3150) during the night. The investigators will collect the SpO2 and pulse rate with this device and then quantify desaturation events.
  The investigators will ask the patient to fill out a questionnaire, which includes the P-SAP score, the STOP-BANG score, the Epworth Sleepiness Scale and the self-reported pain.
  Interventions: Procedure: non-elevated upper body position; Device: Noninvasive wrist pulse oximeter (WristOx Model 3150); Other: Stop-Bang questionnaire; Other: Epworth Sleepiness Scale; Other: P-SAP Score; Other: self-reported pain

INTERVENTIONS:
Procedure: Forty-five degrees elevated upper body position
  Arms: Forty-five degrees elevated upper body position
Procedure: non-elevated upper body position
  Arms: Non-elevated upper body position
Device: Noninvasive wrist pulse oximeter (WristOx Model 3150) — The noninvasive wrist pulse oximeter (WristOx Model 3150) is used to measure the SpO2 and the pulse rate of the patient in the first night after delivery.
Other: Stop-Bang questionnaire — The Stop-Bang questionnaire is a well-established clinical tool to quantify the risk factors of Obstructive Sleep Apnea, which can lead to desaturation in the patient. The STOP Bang questionnaire includes snoring, tiredness, observed apneas, blood pressure, Body Mass Index, age, neck circumference and gender.
  The investigators will ask the patient to answer the questionnaire and measure the neck circumference.
Other: Epworth Sleepiness Scale — The Epworth Sleepiness Scale is a well-established clinical tool to quantify daytime sleepiness. It is clinically used for the diagnosis of sleep disorders.
  The investigators will ask the patient to complete the questionnaire and will specify that the questionnaire pertains to the patient's pre-admission condition.
Other: P-SAP Score — The P-SAP Score is a well-established clinical tool to quantify the risk factors of Obstructive Sleep Apnea, which can lead to desaturation in the patient.
  The investigators will ask the patient to answer the questionnaire and will assess the Mallampati Score. The investigators will also measure the neck circumference and the Thyromental distance.
Other: self-reported pain — A verbal numerical rating scale is used to asses the pain during the study-night.

SUMMARY:
The primary aim of the study is to evaluate the effect of the method of delivery (vaginal delivery vs. cesarean section) on oxygen saturation in the first postpartum night. The investigators hypothesize that nocturnal desaturation occurs more frequently in cesarean section compared with vaginal delivery, expressed as either the duration of SpO2 below 90% or the Oxygen Desaturation Index (ODI). The ODI is defined as number of oxygen desaturations by at least 3 % per hour. Furthermore, the investigators expect a higher pulse rate and a lower mean and minimum SpO2 in the cesarean section group compared with the vaginal delivery group.

The secondary aim of the study is to investigate how the upper body position during sleep (45 degree elevated vs. non-elevated) affects the oxygen saturation during the first postpartum night.

The investigators hypothesize that an upper body elevation to 45 degrees decreases the incidence of desaturation events, expressed as either the duration of SpO2 below 90% or the ODI , compared with a non-elevated body position within each delivery group (vaginal delivery or cesarean section).

The third aim of the study is to identify independent predictors of nocturnal desaturation in postpartum women. To that end, the investigators will administer questionnaires and collect demographic and clinical data according to various obstructive sleep apnea screening scores, including the P-SAP, STOP-Bang, and Epworth Sleepiness Scale. The investigators will also ask the patient to rate the pain during the study night on a verbal numerical rating scale.

DETAILED DESCRIPTION:
Sleep-disordered breathing is common in pregnancy, persisting into the early postpartum period. Postpartum airway obstruction is a main cause of anesthesia-related maternal death in North America. Upper airway edema following labor and delivery may impair pharyngeal anatomy, which can lead to increased vulnerability of the airway collapse during sleep.

This study evaluates whether the kind of delivery (vaginal birth versus cesarean section) has an effect on nocturnal desaturation in the first night after delivery. Furthermore, the investigators examine if the upper body position during sleep has an effect on the occurrence of oxygen desaturation.

In addition, the investigators evaluate if preexisting conditions, as indicated by a high P-SAP or STOP-Bang-score increase the likelihood of nocturnal desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum mothers within 24 hours of delivery
* Age over 18 years.
* Admitted to the Massachusetts General Hospital OB service for the delivery.
* Interventions will be randomly assigned to the patients enrolled in this study

Exclusion Criteria:

* 1 Age under 18 years

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2014-05; Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eikermann, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-elevated Upper Body Position: If the patient is randomized in this study arm after enrollment, the investigators will flatten the patients upper body to a supine position prior to sleeping. The patient will wear a pulseoximeter (WristOx Model 3150) during the night. The investigators will collect the SpO2 and pulse rate with this device and then quantify desaturation events.
  The investigators will ask the patient to fill out a questionnaire, which includes the P-SAP score, the STOP-BANG score, the Epworth Sleepiness Scale and the self-reported pain.
  non-elevated upper body position
  Noninvasive wrist pulse oximeter (WristOx Model 3150): The noninvasive wrist pulse oximeter (WristOx Model 3150) is used to measure the SpO2 and the pulse rate of the patient in the first night after delivery.
  Stop-Bang questionnaire: The Stop-Bang questionnaire is a well-established clinical tool to quantify the risk factors of Obstructive Sleep Apnea, which can lead to desaturation in the patient. The STOP Bang questionnaire
- Forty-five Degrees Elevated Upper Body Position: If the patient is randomized in this study arm after enrollment, the investigators will elevate the patients upper body to 45 degree prior to sleeping. The patient will wear a pulseoximeter (WristOx Model 3150) during the night. The investigators will collect the SpO2 and pulse rate with this device and then quantify desaturation events.
  The investigators will ask the patient to fill out a questionnaire, which includes the P-SAP score, the STOP-BANG score, the Epworth Sleepiness Scale and the self-reported pain.
  Forty-five degrees elevated upper body position
  Noninvasive wrist pulse oximeter (WristOx Model 3150): The noninvasive wrist pulse oximeter (WristOx Model 3150) is used to measure the SpO2 and the pulse rate of the patient in the first night after delivery.
  Stop-Bang questionnaire: The Stop-Bang questionnaire is a well-established clinical tool to quantify the risk factors of Obstructive Sleep Apnea, which can lead to desaturation in the patient.
Period: Overall Study
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
Started | 50 | 49
Completed | 40 | 40
Not Completed | 10 | 9
Not completed — technical issues | 2 | 0
Not completed — participant forgot to wear device | 5 | 5
Not completed — data for less than 60 minutes | 3 | 3
Not completed — participant did not sleep | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (5.5) | 32.5 (5) | 33 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 31 | 32 | 63
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 25 | 32 | 57
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 8 | 3 | 11
Delivery Type [Count of Participants; unit: Participants]
  Vaginal | 20 | 20 | 40
  Cesarean section | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: SpO2 < 90%
Description: Oxygen Saturation (SpO2) value below 90%, assessed by pulse oximetry during the first night after delivery
Time Frame: 48 hours after delivery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
Number analyzed (Participants) | 40 | 40
minutes
  All Types of Delivery | 0.4 [0.0 to 6.4] | 0.0 [0.0 to 0.5]
  Vaginal Delivery | 0.1 [0.0 to 0.3] | 0.0 [0.0 to 0.1]
  Cesarean Section | 4.1 [0.9 to 19.8] | 0.2 [0.0 to 1.8]

2. Secondary Outcome: Oxygen Desaturation Index > 3
Description: ODI (oxygen desaturation index), assessed by pulse oximetry during the first night after delivery. ODI is defined as number of desaturation events per hour; a desaturation event is defined as drop in SpO2 of 3% or more from baseline SpO2. Baseline SpO2 is defined as the mean SpO2 of the SpO2 values taken over the preceding 120 seconds.
Time Frame: 48 hours after delivery
Measure: Median (Inter-Quartile Range); unit: 1/hr
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
Number analyzed (Participants) | 50 | 49
1/hr | 4.0 [2.6 to 6.5] | 3.2 [2.2 to 5.8]

3. Secondary Outcome: Minimal & Mean SpO2
Description: Basic pulseoximetry in the first night after delivery
Time Frame: 48 hours after delivery
Measure: Median (Inter-Quartile Range); unit: percentage of hemoglobin in the blood
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
Number analyzed (Participants) | 40 | 40
percentage of hemoglobin in the blood
  Basal (Mean) SPO2 | 94.7 [93.4 to 95.4] | 95.2 [94.5 to 96.1]
  Nadir (Minimum) SPO2 | 87 [82 to 90] | 90 [87 to 92]

4. Secondary Outcome: P-SAP Score
Description: A Perioperative sleep apnea prediction (P-SAP) Score. This score ranges from 0 to 69, 0 representing low risk of obstructive sleep apnea and 69 representing high risk of obstructive sleep apnea.
Time Frame: 48 hours after delivery
Population: The number analyzed per row differs from the overall number because the analysis was distinguished down by type of delivery and upper body position. Thus, 20 patients belong to each group as seen below.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
Number analyzed (Participants) | 40 | 40
units on a scale
  Vaginal Delivery: number analyzed (Participants) | 20 | 20
  Vaginal Delivery | 1 [1 to 2] | 1 [0 to 2]
  Cesarean Section: number analyzed (Participants) | 20 | 20
  Cesarean Section | 2 [2 to 3] | 2 [1 to 3]

5. Secondary Outcome: STOP-BANG Score
Description: The STOP BANG (This abbreviation consists of the first letter of each question in the questionnaire. S-Snore, T-Tired, O-Observed stop in breathing, P-High blood pressure, B-BMI, A - Age, N-Neck circumference, G-Gender. This questionnaire is a proven tool that can be used to screen for obstructive sleep apnea (OSA). This tool will assess if you are low, moderate or high risk group for sleep apnea. Scores range from 0-8. 0 indicates low risk for sleep apnea, 8 indicates high risk for sleep apnea.
Time Frame: 48 hours after delivery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
Number analyzed (Participants) | 40 | 40
units on a scale
  Vaginal Delivery | 1 [0 to 1] | 1 [0 to 1]
  Cesarean Section | 1 [1 to 2] | 2 [1 to 2]

6. Secondary Outcome: Pain-score on a Verbal Numerical Rating Scale
Description: Assessment of intensity of acute pain. Measured from 0-10, 0 being no pain and 10 being highest level of pain.
Time Frame: 48 hours after delivery
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
Number analyzed (Participants) | 40 | 40
units on a scale
  Vaginal Delivery | 3 [1 to 4] | 3 [2 to 5]
  Cesarean Section | 4 [2 to 6] | 4 [3 to 6]

7. Secondary Outcome: Average Pulse Rate
Description: As measured in beats per minute
Time Frame: 48 Hours after delivery
Measure: Median (Inter-Quartile Range); unit: beats per minute
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
Number analyzed (Participants) | 40 | 40
beats per minute | 78.8 [69.9 to 86.1] | 75.2 [68.6 to 87.3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected 48 hours after delivery.
Arm/Group | Non-elevated Upper Body Position | Forty-five Degrees Elevated Upper Body Position
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 0/50 | 0/49

LIMITATIONS AND CAVEATS:
The true prevalence of pregnancy-associated OSA is unknown in our cohort due to lack of diagnosis by polysomnography. We obtained questionnaires validated as OSA screening tools, but their ability to predict OSA in pregnancy remains controversial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT02330055/SAP_000.pdf
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT02330055/Prot_001.pdf